CLINICAL TRIAL: NCT05724992
Title: Standardised Genetic Profiling of Subjects Belonging to the Italian Multicenter Registry of Prospective Surveillance of Subjects at Genetic Risk of Pancreatic Cancer
Brief Title: Familial Pancreatic Cancer PROPHilation Program in Italy
Acronym: PROPH-ITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Associazione Italiana per lo Studio del Pancreas (Other)
Collaborators: General and Pancreatic Surgery Unit, University of Verona (Unknown); Fondazione Valsecchi (Unknown); Associazione Oltre La Ricerca (Unknown); Genomica srl (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROPH-ITA
Record Dates: First submitted 2022-12-20; First posted 2023-02-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Candidates for Hereditary Pancreatic Cancer Testing
Keywords: Pancreatic Cancer; Pancreatic Cancer familiarity; Genetic profiling; Genetic predisposition; Pancreatic Cancer surveillance
MeSH Terms: conditions — Pancreatic Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saliva testing swab (Other): Subjects with familiarity with pancreatic cancer enrolled into the IRFARPC registry (NCT04095195) will be submitted to buccal swab for saliva-based genetic testing
  Interventions: Genetic: Saliva swab testing

INTERVENTIONS:
Genetic: Saliva swab testing — 41 pancreatic cancer predisposition genes will be tested through a saliva-based swab

SUMMARY:
The goal of the PROPH-ITA Study is to perform genetic testing in family members of pancreatic cancer patients who may have a genetic predisposition. The subjects belong to the Italian Registry of Families At Risk of Pancreatic Cancer (IRFARPC, #NCT04095195). This investigational study will assess the genetic background of subjects with familiarity with pancreatic cancer only.

Participants may accept to undergo genetic testing as part of the IRFARPC registry, through a saliva-swab-based 41-gene panel test.

Up to 3,000 participants will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled on the IRFARPC registry
* Having familiarity for pancreatic cancer (according to the IRFARPC criteria, Capurso et al. Dig Liv Dis, 2020)
* Willingness to participate in saliva-swab-based genetic testing

Exclusion Criteria:

- Already known genetic mutation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Presence - absence of predisposing mutations | 5 years
  Prevalence of genetic mutations over the total tested

SECONDARY OUTCOMES:
Correlation of genetic mutations with personal oncological history | 5 years
  Correlation between presence of predisposing mutation and prevalence of cancers
Correlation of genetic mutations with familial oncological history | 5 years
  Correlation between presence of predisposing mutation and prevalence of cancers in the family

CONTACTS AND LOCATIONS:
Locations (1):
- Chirurgia generale e del Pancreas Azienda Ospedaliera Universitaria Integrata, Verona, Italy

IPD SHARING:
Plan to Share IPD: No